CLINICAL TRIAL: NCT00211328
Title: Treatment of Idiopathic Perifoveal Telangiectasia (IPT) With Open-Label Anecortave Acetate (15mg.).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Manhattan Eye, Ear & Throat Hospital (Other)
Collaborators: Alcon Research (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AA in IPT
Expanded Access: Available
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Idiopathic Perifoveal Telangiectasia
MeSH Terms: interventions — anecortave acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: anecortave acetate

SUMMARY:
Idiopathic Perifoveal telangiectasia is a poorly understood disorder that involves the growth of blood vessels around the center of the macula(perifoveal region). These blood vessels may extrend beneath the retina to produce an area of sub-retinal neosvascularization(growth of abnormal blood vessels under the retina which "leak" fluid, causing reduction in vision. Limited forms of treatment are available in managing the neovascularization and its consequences. Anecortave Acetate injection is considered as an attempt to control the growth of the abnormal blood vessels.

DETAILED DESCRIPTION:
In this open-label pilot study, an initial patient, which presented with IPT and SRN, was treated with promising success and five additional patients were then recruited. So this is a report on six eyes of the first six patients with this disease who presented in our practice. The Food and Drug Administration (FDA) granted our site permission to enroll these patients. While anecortave acetate has not yet been approved by the FDA, it has been used in phase 2/3 trials for the treatment of AMD. An informed consent was obtained from each patient. IRB approval was obtained from Manhattan Eye, Ear, and Throat Hospital.

Patients received a posterior juxtascleral injection of 15 mg of anecortave acetate delivered adjacent to the macula using the specially designed curved cannula by Alcon, Inc. Visual acuity (VA) and intraocular pressure (IOP) were measured on each study visit. Fluorescein angiography was used to complement the standard clinical biomicroscopic examination of the macula at baseline and at 3 months intervals. On the first day post-injection, patients had an additional ophthalmic examination including VA testing, biomicroscopy, and IOP measurement.

A 6-month retreatment interval was established for this study based on laboratory data demonstrating that anecortave acetate administered as a slow-release depot adjacent to the posterior scleral surface provided therapeutic drug levels in the adjacent choroid and retina for up to 6 months (9). If patients were clinically unstable or unimproved six months after enrollment, they were offered thermal laser treatment or photodynamic therapy (PDT) in conjunction with the anecortave acetate injection. Patients who were unstable as early as 3 months after enrollment were offered the option to be treated with either thermal laser or PDT. This did not disqualify them from being eligible for the repeat anecortave acetate injection at month 6.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of patients with Idiopathic Perifoveal Telangiectasia(IPT).
2. Patients must be 18 years of age or older to receive treatment.
3. Visual acuity of 20/30 to 20/320 Study Eye on the ETDRS visual acuity chart.
4. Visual acuity of 20/800 or better Fellow Eye on the ETDRS visual acuity chart .

Exclusion Criteria:

1. Patient with significantly compromised visual acuity in the study eye due to concomitant ocular conditions.
2. Patients who have undergone intraocular surgery within last 2 months.
3. Patient participating in any other investigational drug study.

3.Use of an investigational drug or treatment related or unrelated to their condition within 30 days prior to receipt of study medication.

4.Inability to obtain photographs to document CNV (including difficulty with venous access).

5.Patient with significant liver disease or uremia. 6.Patient with known adverse reaction to fluorescein and indocyanine green or iodine.

7.Patient has a history of any medical condition which would preclude scheduled visits or completion of study.

8.Patient has had insertion of scleral buckle in the study eye. 9.Patient has received radiation treatment 10.Patient is on anticoagulant therapy with the exception of aspirin 11.Patient is pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2002-03; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
To investigate the use of anecortave acetate fot treatment of idiopathic perifoveal telangiectasia | 24 months

SECONDARY OUTCOMES:
mean change of VA (ETDRS)from baseline to 24 months | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A. Yannuzzi, MD, Principal Investigator — Manhattan Eye, Ear & Throat Hospital
Locations (1):
- Manhattan Eye, Ear & Throat Hospital, New York, New York, United States